CLINICAL TRIAL: NCT05556811
Title: Evaluation of Specific Light Algorithms to Maintain and Restore Circadian Melatonin Rhythmicity in Critically Ill Patients
Brief Title: HEaling LIght Algorithms for the ICU Patient
Acronym: HELIA-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Alawi Luetz, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20018170
Record Dates: First submitted 2022-08-18; First posted 2022-09-27 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Critical Care; Phototherapy
Keywords: Light therapy; Melatonin; Critical Care; Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LSA-1 (Active Comparator): Light Scheduling Algorithm-1 (LSA-1): High circadian effective irradiances + Blue Enriched Light episodes
  Interventions: Device: Dynamic Light Therapy Device, LSA-1
- LSA-2 (Active Comparator): Light Scheduling Algorithm-2 (LSA-2): High circadian effective irradiances without Blue Enriched Light episodes.
  Interventions: Device: Dynamic Light Therapy Device, LSA-2
- LSA-3 (Active Comparator): Light Scheduling Algorithm-3 (LSA-3): Irradiance levels comparable to conventional hospital lighting (control group).
  Interventions: Device: Dynamic Light Therapy Device, LSA, 3

INTERVENTIONS:
Device: Dynamic Light Therapy Device, LSA-1 — Dynamic Light Therapy
  Arms: LSA-1
Device: Dynamic Light Therapy Device, LSA-2 — Dynamic Light Therapy
  Arms: LSA-2
Device: Dynamic Light Therapy Device, LSA, 3 — Dynamic Light Therapy
  Arms: LSA-3

SUMMARY:
The purpose of this prospective, randomized controlled trial is to investigate if mechanically ventilated patients who are treated with a Light Scheduling Algorithm with high circadian effective irradiances are better able to preserve and induce physiological melatonin rhythms compared to patients who are treated with an application of lower irradiances.

The investigators will further evaluate the impact on delirium prevalence, stress level and general outcome parameters.

DETAILED DESCRIPTION:
Circadian disruption affects the majority of ICU patients and has far-reaching effects on organ functioning. At the level of the central nervous system, circadian misalignment facilitates executive cognitive dysfunction and the development of brain disorders such as ICU delirium.

The suprachiasmatic nucleus (SCN) in the hypothalamus serves as the master pacemaker that sets the timing of circadian rhythms by regulating neuronal activity. Its function is determined by environmental factors, especially visible light with a high content of blue light components. Light as a photoperiodic signal has a great impact on the regulation of the epiphyseal melatonin secretion and the entrainment of the day-night rhythm. As a result using light therapy to maintain or entrain circadian rhythm seems to be a promising approach to prevent delirium in critically ill patients. The specific light effect on the rhythmicity of the melatonin levels is to be examined in a randomized controlled study design, which includes the application of three different Light Scheduling Algorithms. In this context a highly specialized light ceiling was installed in two patient treatment rooms. A Light Scheduling Algorithm (LSA) consists of specified values for illuminance [lux] and correlated color temperature (CCT, [kelvin]) for different time points and durations within a 24-hour period. These values are calculated by assessment of photometric light measures with regard to visual light effects as well as non-image-forming functions at the patients bedside.

Patients will be randomly allocated in to 3 treatment groups: (1) LSA-1 (high circadian effective irradiances + blue Light Intervention), (2) LSA-2 (high circadian effective irradiances without blue light intervention) and (3) LSA-3 (standard irradiances, Control Group). All LSAs will be applied to the patient using VitalSky Advanced. For the purpose of validation of efficacy of specific light interventions, blood samples for measurement of melatonin concentration will be collected.

The temporal study sequence is defined by treatment days and measurement series periods (SMAP-1 to SMAP-4, Serum Melatonin Assessment Period). SMAP-1 starts on the first morning at 06:00 a.m. after study inclusion. SMAP-1 through SMAP-4 each define 24-hour periods in which the blood melatonin concentration is determined every 4 hours (6 am, 10 am, 2 pm, 6 pm, 10 pm, 2 am, 6 am). The SMAP-1 is intended to determine the patient's individual melatonin baseline. SMAP-2 to SMAP-4 start only when the patient has reached a stable level of wakefulness (RASS ≥-3 ). It can be assumed that the light intervention will only have an effect on melatonin balance from this level of wakefulness. A total of 4 SMAPs are planned per study patient.

Main Hypothesis:

Ventilated ICU patients receiving increased irradiance lighting may differ in the rhythmicity of serum melatonin concentrations and more frequently exhibit physiologic circadian melatonin secretions compared with patients receiving conventional irradiance lighting.

Secondary Hypotheses:

1. Ventilated intensive care patients receiving illumination with increased irradiance and phases of Blue-Enriched White light (BEW) differ in the rhythmicity of serum melatonin concentrations compared with patients receiving illumination with increased irradiance but without BEW.
2. Ventilated intensive care patients receiving illumination with increased irradiance and phases with BEW differ in the rhythmicity of serum melatonin concentrations compared with patients receiving illumination with conventional irradiance.
3. Ventilated intensive care patients receiving illumination with increased irradiance without phases with BEW differ in the rhythmicity of serum melatonin concentrations compared with patients receiving illumination with conventional irradiance.
4. Ventilated intensive care patients receiving increased irradiance lighting and periods of BEW have a lower incidence of delirium than patients receiving conventional irradiance lighting.
5. Ventilated intensive care patients receiving increased irradiance lighting and periods of BEW have lower delirium severity than patients receiving conventional irradiance lighting.

ELIGIBILITY:
Inclusion Criteria:

* Patient capable of giving consent or additionally existing legal caregiver/authorized representative in case of non-consenting patients in the intensive care unit
* Male and female patients with age ≥ 18 years
* Expected intensive care unit stay ≥ 5 days
* Invasive mechanical ventilation or non-invasive mechanical ventilation (with positive ventilation pressure > 6 hours/day or high flow >30 liters) on the day of ICU admission

Exclusion Criteria:

* Participation in other clinical studies during the study period and ten days before
* Patients with psychiatric diseases
* Patients with a history of stroke and known severe residual cognitive deficits
* Patients with a history of cardiopulmonary arrest or pulseless electric activity with cardiopulmonary resuscitation followed by therapeutic hypothermia during entire hospital stay
* Analphabetism
* Anacusis or Hypoacusis with hearing aid device, Amaurosis
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* History of sleep-related breathing disorders
* History or suspicion of hypoxic brain damage
* History or suspicion of elevated intracranial pressure in the last 7 days before study inclusion
* Patients with an open chest after cardiac surgery
* Patient has a power of attorney or patient's provision, where he/she refuses participation in any clinical trial
* The informed consent of the patient or the subject's legally acceptable representative can't be obtained in time
* Severe eye diseases
* History of photoallergic reactions
* History of visually triggered seizures

Termination criteria:

Under the following conditions, premature withdrawal of a Patient from the study according to the termination criteria will occur:

* Personal request of the patient/caregiver/authorized representative.
* Any other situation in which, in the opinion of the study physician, continued participation in the clinical trial is not in the best interest of the of the patient
* Subsequent occurrence of an exclusion criterion

Premature termination of the study or discontinuation of the entire study may be considered because of the following circumstances:

* Decision of the principal investigator in case of unacceptable risks under Benefit-risk consideration
* New (scientific) findings during the term of the clinical study that may compromise the safety of the study participants (positive risk-benefit balance no longer given).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in serum melatonin concentration | Plasma melatonin levels will be assessed for a maximum of five 24-hour periods. Blood samples will be collected every 4 hours within each series of measurements. (6am, 10am, 2pm, 6pm, 10pm, 2am, 6am).
  Prevalence of physiological circadian rhythmicity measured by serum melatonin concentrations

SECONDARY OUTCOMES:
Prevalence of intensive care unit delirium | Participants will be followed up to 6 days after intensive care unit admission
  Delirium will be measured with the Confusion Assessment Method for the intensive care unit (CAM-ICU), Binary scale (Positive/Negative)
Delirium Severity | Participants will be followed up to 6 days after intensive care unit admission
  Delirium Severity will be measured with the Intensive Care Delirium Screening Checklist (ICDSC). The higher the score the worse - higher score = higher delirium severity(ICDSC)
Depth of Sedation | Participants will be followed up to 6 days after intensive care unit admission
  Level of sedation will be measured with the Richmond Agitation-Sedation-Scale (RASS), -5 to +4, negative scores translates to a higher degree of sedation.
Severity of Pain | Participants will be followed up to 6 days after intensive care unit admission
  Severity of pain will be measured with the Numeric Rating Scale (NRS), or the Visualized Numeric Rating Scale (NRS-V) or the Faces Pain Scale-Revised (FPS-R) or the Behavioral Pain Scale (BPS) or the Behavioral Pain Scale for Non- Intubated (BPS-NI). A higher score corresponds to a higher severity of pain.Score values from 0 to 10. A higher score means worse outcome
Patient comfort | Participants will be followed up to 6 days after intensive care unit admission
  Distress thermometer
Duration of mechanical and non-mechanical ventilation | Participants will be followed up until ICU discharge
  Hours
ICU length of stay | Participants will be followed up until ICU discharge
  Days
Hospital length of stay | Participants will be followed up until hospital discharge
  days
Sepsis | Participants will be followed up to 6 days after intensive care unit admission
  Does patient fulfil sepsis criteria (Yes/No)
Septic Shock | Participants will be followed up to 6 days after intensive care unit admission
  Does patient fulfil criteria for septic shock (Yes/No)
Sequential Organ Failure Assessment (SOFA-Score) | Participants will be followed up to 6 days after intensive care unit admission
  Predicts ICU mortality based on lab results and clinical data.
Simplified Acute Physiology Score (SAPS II) | Participants will be followed up to 6 days after intensive care unit admission
  Estimates mortality in ICU patients, comparable to APACHE II.
Therapeutic Intervention Scoring System (TISS-28) | Participants will be followed up to 6 days after intensive care unit admission
  The Simplified Therapeutic Intervention Scoring System TISS-28 consists of 28 items. It is intended to accurately measure the level of care required for a patient in the Intensive Care Unit (ICU)
Acute Physiological and Chronic Health Evaluation 2 Score (APACHE II) | Participants will be followed up to 6 days after intensive care unit admission
  The Acute Physiology and Chronic Health Evaluation (APACHE II) is a severity score and mortality estimation tool developed from a large sample of ICU patients in the United States.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of Research Group — https://cociwg.org
- See also: Website of Department — https://anaesthesieintensivmedizin.charite.de/en/